CLINICAL TRIAL: NCT01820039
Title: FertiScreen: an Online Application to Improve the Quality of Fertility Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FertiScreen
Record Dates: First submitted 2013-03-14; First posted 2013-03-28 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-03

CONDITIONS: Unexplained Subfertile Couples With a Good Prognosis.
Keywords: e-health intervention; infertility; primary care; referral rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FertiScreen (Experimental): all patients between 18 and 38 years, consulting their general practitioner for infertility will be asked to use FertiScreen.
  Interventions: Other: FertiScreen

INTERVENTIONS:
Other: FertiScreen — FertiScreen is an online application to assess whether referral is necessary or expectant management is indicated.

SUMMARY:
Objectives The investigators present an online application to empower and inform patients and improve guideline adherence in unexplained subfertility. Thereby the investigators expect to reduce overtreatment in fertility care with higher quality of care.

Methods The investigators conduct a prospective cohort study including couples with a diagnosis of unexplained subfertility. Couples consulting their general practitioner with an unfulfilled child wish will be offered to use FertiScreen. FertiScreen is an online application, in which patients are asked questions about their fertility problem (ie menstrual cycle, age, duration of child wish and the results of the Chlamydia Trachomatis antibody titre and semen analysis). FertiScreen then uses the validated prediction model of Hunault to calculate couples' chance of natural conception during the next twelve months. In addition, patients can find links to extra information concerning subfertility. Couples can then initiate an online consultation with their general practitioner and a gynaecologist, in order to discuss their results and prognosis. When the calculated prognosis of spontaneous conception within one year is >30%, tailored expectant management for 6-12 months will be advised, as no benefit can be expected from fertility treatment.

Questionnaires will be sent to patients as well as to their caregivers (general practitioner, gynaecologist). These questionnaires will focus on the use of FertiScreen (System Usability Scale) and the different domains of quality of care (effectiveness, cost-effectiveness, safety, patient-centredness). For the latter, the investigators use the Hospital Anxiety and Depression Scale and the Patient Centredness Questionnaire for Infertility.

In order to be able to draw conclusions, the investigators will conduct a baseline measurement among couples with unexplained subfertility who have been referred to a fertility clinic. Their data will be abstracted from their medical records and they will receive the aforementioned questionnaires as well (except for the System Usability Scale).

The investigators will recruit couples presenting to general practitioners in the Nijmegen area (which for second line treatment consists of one general hospital and one academic hospital). To detect an increase in guideline adherence of the current 60% to 75% with a power of 80% (P<0,05), the investigators need to include 152 couples in the before as well as in the after measurement.

ELIGIBILITY:
Inclusion Criteria:

* couple consulting their general practitioner with subfertility
* women >18 years and <38 years
* one of the partners Dutch speaking
* access to the Internet
* residing in the Netherlands
* unfulfilled childwish for at least 6 months

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the application: adherence to tailored expectant management | Two years
  The adherence to tailored expectant management: measured by the percentage of patients with unexplained infertility with a good prognosis of spontaneous conception within one year (>30%) with tailored expectant management.

SECONDARY OUTCOMES:
experiences with FertiScreen | two years
  Among the patients the focus will be on ease of use, speed of use, sense of privacy, the extent to which the experience meet previous expectations and the recognisability of the given advise. Among health care providers, the evaluation will focus on the experienced changes in the daily care.

OTHER OUTCOMES:
effects on quality of care | two years
  Efficiency: economic analysis (number of consultations in the second line and the number of diagnostic tests carried out.
  Safety: we will measure complaints of anxiety and depression and quality of life at a patient level.
  Future implications: we will give advises for implementation strategy to optimize use of FertiScreen.

CONTACTS AND LOCATIONS:
Overall Officials: Jan AM Kremer, MD, PhD, Study Director — IQ Healthcare, UMC St Radboud, Nijmegen, The Netherlands
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, PO Box 9101, Netherlands